CLINICAL TRIAL: NCT05050890
Title: Prognostic Value of Circulating Tumor DNA Dosing in Patients in Neoadjuvant Breast Neoplasia
Acronym: GIRO_ctDNA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Principal Investigator, Camila Giro, Principal Investigator, Instituto Brasileiro de Controle do Cancer
Other Study IDs: 32158620.0.0000.0072
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-08

CONDITIONS: Breast Neoplasm
Keywords: Breast Cancer; Liquid Biopsy; ctDNA; Pathologic complete response
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer: Breast cancer patients who are currently receiving neoadjuvant therapy
  Interventions: Other: ctDNA level during neoadjuvant chemotherapy

INTERVENTIONS:
Other: ctDNA level during neoadjuvant chemotherapy — ctDNA samples will be collected from patients at baseline, during neoadjuvant therapy (every 15 days) and before the surgical procedure

SUMMARY:
This is a cohort, single-center, prospective study that seeks to analyze the circulating tumor DNA (ctDNA) in patients diagnosed with breast cancer, who will undergo neoadjuvant treatment.

DETAILED DESCRIPTION:
Breast cancer is a major public health problem, being the most common cancer in women worldwide. Breast cancer can be diagnosed through multiple tests, including an imaging and tissue biopsy. However, accurate assessment and prediction of the response is a major challenge. Circulating tumor DNA (ctDNA) has shown promise in the detection of breast cancer and clinical and cancer outcomes.

This study aims to evaluate a possible correlations between ctDNA levels with the pathological complete response and detection of residual disease after neoadjuvant therapy in patients with breast cancer.

In order to start ctDNA surveillance, patients will be asked to participate in blood draws, every 15 days, during neoadjuvant standard institutional treatment and allow study staff to review medical records.

ELIGIBILITY:
Inclusion Criteria:

* Information to the patient and signed informed consent;
* Locally advanced breast cancer that is a candidate for neoadjuvant therapy;
* Histological diagnosis of localized invasive breast carcinoma, confirmed by the pathologist, with or without expression of hormone receptors, and/or with the presence of HER-2.

Exclusion Criteria:

* Metastatic breast cancer (Stage IV);
* Additional invasive malignant disease;
* Known psychiatric or substance abuse disorders that may interfere with cooperation with study requirements;
* Presents any organic condition that makes it impossible to carry out chemotherapy treatment;
* Pregnant or lactating women
* Received previous treatment for breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer who are considered possible candidates for neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
The concentration of circulating DNA(ctDNA) | From date of enrollment until the date of end of neoadjuvant treatment, assessed up to 6-7 months
  Circulating tumor DNA (ctDNA) levels will be measured each 15 days until end of neoadjuvant therapy, through peripheral blood collection

SECONDARY OUTCOMES:
Change from baseline ctDNA alterations to end of neoadjuvant treatment | Up to approximately 7 months starting from Baseline until end of neoadjuvant treatment
  The percentage of patients with ctDNA alterations will be provided over time of neoadjuvant treatment to characterize the biological evolution of the disease in each patient. The association of these alterations with clinical outcomes will also be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Camila Giro, MD, Principal Investigator — IBCC Oncologia
Locations (1):
- IBCC Oncologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The findings will be shared and discussed with all investigators in the study. A study manuscript, having received contributions from all authors, will be submitted for publication in scientific circles.